CLINICAL TRIAL: NCT03761186
Title: DANCE (Diabetes ANd CarbohydratEs). Does the Amount of Dietary Carbohydrates Affect Insulin Requirements and Metabolic Control in Type 1 Diabetes? Comparative Study of Traditional Diabetes, Moderately Low and Strictly Low Carbohydrate Diet
Brief Title: Comparison of Low, Moderate and High Carbohydrate Diet on Insulin Requirements and Metabolic Control in Type 1 Diabetes
Acronym: DANCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Anneli Björklund (Other)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Sponsor-Investigator, Anneli Björklund, Principal Investigator, Senior Consultant, Associate Professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2018/218-31
Record Dates: First submitted 2018-11-26; First posted 2018-12-03 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Type1diabetes
Keywords: type 1 diabetes; low carbohydrate diet; randomized trial; adults; insulin; metabolic control
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Nurses that will take lab samples as well as laboratory personal that analyses the samples will be masked. Due to the nature of the study, it is not possible to mask the participants or the care providers/investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- traditional diabetes diet (Active Comparator): Participants in this arm will follow a diet with carbohydrate intake 50-60% of total energy intake
  Interventions: Behavioral: traditional diabetes diet
- moderately low carbohydrate diet (Experimental): Participants in this arm will follow a diet with carbohydrate intake 30-40% of total energy intake
  Interventions: Behavioral: moderately low carbohydrate diet
- strictly low carbohydrate diet (Experimental): Participants in this arm will follow a diet with carbohydrate intake 15-20% of total energy intake
  Interventions: Behavioral: strictly low carbohydrate diet

INTERVENTIONS:
Behavioral: traditional diabetes diet — Diet with carbohydrate content 50-60% of total energy intake
  Arms: traditional diabetes diet
Behavioral: moderately low carbohydrate diet — Diet with carbohydrate content 30-40% of total energy intake
  Arms: moderately low carbohydrate diet
Behavioral: strictly low carbohydrate diet — Diet with carbohydrate content 15-20% of total energy intake
  Arms: strictly low carbohydrate diet

SUMMARY:
The scientific basis for dietary recommendations in type 1 diabetes is almost lacking, with the current recommendations being based on type 2 diabetes studies. Therefore the overall purpose of this study is to improve the current evidence for dietary recommendations to people with type 1 diabetes.

Study aim: To compare how a strictly low carbohydrate diet, a moderately low carbohydrate diet and a traditional diabetes diet (with higher amounts of carbohydrates) affect insulin requirements and metabolic control in individuals with type 1 diabetes.

Carbohydrate intake is 50-60% of the total energy intake in the traditional diabetes diet, 30-40% in the moderately low carbohydrate diet and 15-20% in the strictly low carbohydrate diet with a minimum of 50 g carbohydrates/day. A diet with less than 50 g carbohydrates/day is usually called very low carbohydrate diet or ketogenic and will not be tested in this study.

Those who wish to participate and meet the inclusion criteria (and none of the exclusion criteria) will be randomized to one of the three diets. The duration of the intervention is 6 months after which the participants will be able to choose their own diet for another 6 months. The main study visits are at baseline (screening and study start), 3, 6, 9, and 12 months. Shorter visits will be at 3 and 6 weeks. The participants will meet with a study nurse, dietitian and doctor. They will attend two carbohydrate counting courses before the start of the intervention in order to be able to match their insulin to the amount carbohydrates they eat. Participants will receive written materials about their diets with menus and recipes for better adherence to the diet.

The primary endpoint is the change in insulin requirements within and between groups (for secondary endpoints please see relevant section). For assessing the different endpoints the participants will provide blood, urine and feces samples for lab analyses as well as register their insulin use, blood glucose, diet, physical activity and any blood ketones or hypoglycemia electronically or in written forms. Continuous/flash glucose monitoring (CGM/FGM) will be also used. Dietary assessment and adherence will be based on 3-4 day food diaries before every scheduled study visit.

ELIGIBILITY:
Inclusion Criteria:

* To have had type 1 diabetes for at least 1 year
* Age >=20 years old

Exclusion Criteria:

* Cardiovascular disease NYHA class IIIB or more
* Kidney disease > stadium 3
* Liver disease, alanine aminotransferase (ALAT) ≥ 2 µkat/L,
* BMI < 18.5 kg/m^2
* c-peptide ≥ 0.3 nmol/l
* Pregnant/breastfeeding women, women that plan to get pregnant during study period
* Other circumstances, which, according to the examiner, make it difficult for an individual to participate.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Change in insulin use | screening, day 0, 3 weeks, 6 weeks, 3 months, 6 months, 9 months, 12 months
  measured in international units (IU) and percentage.

SECONDARY OUTCOMES:
Change in HbA1c | screening, 3 weeks, 6 weeks, 3 months, 6 months, 9 months, 12 months
  mmol/mol
Change in concentration of total cholesterol | screening, 3 months, 6 months, 9 months, 12 months
  mmol/L
Change in concentration of triglycerides | screening, 3 months, 6 months, 9 months, 12 months
  mmol/L
Change in concentration of HDL-cholesterol | screening, 3 months, 6 months, 9 months, 12 months
  mmol/L
Change in concentration of LDL-cholesterol | screening, 3 months, 6 months, 9 months, 12 months
  mmol/L
Ratio of LDL/HDL | screening, 3 months, 6 months, 9 months, 12 months
  absolute number
Concentration of glucagon | screening, 3 months, 6 months, 9 months, 12 months
  pmol/L
Change in markers of glycemic variability (TIR, TAR, TBR, mean sensor glucose with SD, CV) | screening, 3 months, 6 months, 9 months, 12 months
  mmol/L
Change in weight | screening, 3 weeks, 6 weeks, 3 months, 6 months, 9 months, 12 months
  kg
Change in BMI | screening, 3 weeks, 6 weeks, 3 months, 6 months, 9 months, 12 months
  kg/m^2
Change in abdominal circumference | screening, 3 weeks, 6 weeks, 3 months, 6 months, 9 months, 12 months
  cm
Change in concentration of p-creatinine | screening, 3 months, 6 months, 9 months, 12 months
  micromol/L
Change in estimated Glomerular Filtration Rate (eGFR) | screening, 3 months, 6 months, 9 months, 12 months
  mL/min/1,73 m2
Change in microalbuminuria | screening, 3 months, 6 months, 9 months, 12 months
  morning U-Alb/Crea (mg/mmol)
Concentration of Insulin-like Growth Factor 1 (IGF-I) | screening, 3 months, 6 months, 9 months, 12 months
  microg/L
Concentration of Insulin-like Growth Factor - binding protein 1 (IGFBP-1) | screening, 3 months, 6 months, 9 months, 12 months
  microg/L
Concentration of leptin | screening, 3 months, 6 months, 9 months, 12 months
  microg/L
Concentration of adiponectin | screening, 3 months, 6 months, 9 months, 12 months
  mg/L
Concentration of interleukin 6 (IL-6) | screening, 3 months, 6 months, 9 months, 12 months
  ng/L
Concentration of high sensitivity c-Reactive Protein (Hs-CRP) | screening, 3 months, 6 months, 9 months, 12 months
  mg/L
Measurement of lipopolysaccharides (LPS) activity using the Limulus Amebocyte Lysate (LAL) assay | screening, 3 months, 6 months, 9 months, 12 months
  measured in endotoxin units (EU)/ml
Concentration of glutaredoxin 1 (GRX-1) | screening, 3 months, 6 months, 9 months, 12 months
Concentration of Oxidized LDL | screening, 3 months, 6 months, 9 months, 12 months
Total Antioxidant Capacity (TAC) | screening, 3 months, 6 months, 9 months, 12 months
Concentration of reactive oxygen species (ROS) | screening, 3 months, 6 months, 9 months, 12 months
Plasma metabolites assessed by untargeted liquid chromatography - mass spectrometry (LC-MS) metabolomics | screening, 3 months, 6 months, 9 months, 12 months
Score from the Short Form 36 (SF-36) questionnaire | screening, 3 weeks, 6 weeks, 3 months, 6 months, 9 months, 12 months
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health.The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Score from the Well-being Questionnaire-12 (WBQ-12) | screening, 3 weeks, 6 weeks, 3 months, 6 months, 9 months, 12 months
  This questionnaire is designed to measure general well-being, including negative well-being, energy and positive well-being. The negative well-being scale score (range 0-12) is reversed and then summed with the Energy score (range 0-12) and Positive score (range 0-12) to produce a general well-being score (range 0-36). The higher the score the greater the sense of general well-being.
Score from the Diabetes Treatment Satisfaction Questionnaire (DTSQ) | screening, 3 weeks, 6 weeks, 3 months, 6 months, 9 months, 12 months
  The DTSQ has been developed to assess patient satisfaction with diabetes treatment. The questionnaire is composed of two different factors. The ﬁrst factor assesses treatment satisfaction and consists of six questions and the second factor consists of two questions, which assess the burden from hyper- and hypoglycemia. Treatment satisfaction is assessed as the sum of the scores of the six questions on the ﬁrst factor (total score 36), with a higher score indicating higher treatment satisfaction.
Time taken to complete the Trail making test A+B | screening, 3 weeks, 6 weeks, 3 months, 6 months, 9 months, 12 months
  The Trail Making Test is a neuropsychological test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. The time taken to complete the test is used as the primary performance metric, measured in seconds and or minutes.

OTHER OUTCOMES:
Carbohydrate intake | screening, 3 weeks, 6 weeks, 3 months, 6 months, 9 months, 12 months
  in grams/day
Energy intake from carbohydrates | screening, 3 weeks, 6 weeks, 3 months, 6 months, 9 months, 12 months
  % of total energy intake
Daily energy intake of participants | screening, 3 weeks, 6 weeks, 3 months, 6 months, 9 months, 12 months
  kcal/day
Frequency of intake of different foods measured by a Food frequency questionnaire (FFQ) | screening, 6 months,12 months
  The participants will fill in how frequent they consume 132 different food items. The available frequency responses are: 0/month, 1-3/month, 1-2/week, 3-4/week, 5-6/week, 1/day, 2/day, 3+/day.

CONTACTS AND LOCATIONS:
Overall Officials: Anneli Björklund, MD, PhD, Principal Investigator — Department of Endocrinology at Karolinska University Hospital and Academic Specialistcentrum
Locations (1):
- Center for Diabetes, Academic Specialistcenter, Stockholm, Sweden